CLINICAL TRIAL: NCT03679286
Title: Comparative Analysis of the Entegrion Point of Care Coagulation Monitor (PCM) With ROTEM in the Measurement of Viscoelastic Coagulation Parameters
Brief Title: Comparative Analysis of PCM With ROTEM in the Measurement of Viscoelastic Coagulation Parameters
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Entegrion, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PCM-002
Record Dates: First submitted 2018-08-30; First posted 2018-09-20 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Hemostasis Monitoring
Keywords: Coagulation
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All subjects: No intervention
  Interventions: Device: PCM and ROTEM

INTERVENTIONS:
Device: PCM and ROTEM — Test of blood sample by both PCM and ROTEM

SUMMARY:
To determine if PMC viscoelastic coagulation parameters correlate with those generated by a marketed device in adult patients who require hemostasis monitoring or who are at risk of bleeding or thrombotic indications

DETAILED DESCRIPTION:
The primary aim of this study is a performance evaluation of the PCM coagulation monitor in comparison to the ROTEM thromboelastometry system.

To include a measurement of the entire range of the test system, subjects with a medical management need that requires the measurement of their hemostasis status (such as PT/PTT, INR) or are at risk for being hypo-coagulable or hyper-coagulable will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* In opinion of investigator, absence of anything that precludes subject from being good study candidate
* Informed consent
* Order for measurement of hemostasis status of patients who are at risk for being hyper-coagulable or hypo-coagulable due to clinical diagnosis or medical need

Exclusion Criteria:

* Previous enrollment in study
* Incarcerated
* Heparin infusion in prior 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients who have a medical management need that requires measurement of their hemostasis status or are at risk of being hypocoagulable or hypercoagulable
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-08-20 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Method comparison: Deming regression analysis (PCM and ROTEM NATEM) | Parameter differences assessed at time of blood sampling
  Deming regression will be used to compare the PCM and the ROTEM NATEM assay (which reports clotting time, speed of clot formation, maximal clot firmness and clot lysis)

SECONDARY OUTCOMES:
Method comparison: Deming regression analysis (PCM and ROTEM INTEM, EXTEM) | Parameter differences assessed at time of blood sampling
  Deming regression will be used to compare the PCM and the ROTEM INTEM and EXTEM assays (which both report clotting time, speed of clot formation, maximal clot firmness and clot lysis)
Correlation between abnormalities | Parameter differences assessed at time of blood sampling
  Correlation between abnormalities as assessed by conventional coagulation assays (such as fibrinogen concentration, CBC, PT, PTT, INR), vital signs, demographics or trauma (if any)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Washington University in St. Louis, St Louis, Missouri
  - Ohio State University, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania